CLINICAL TRIAL: NCT00469742
Title: Safety Profile of Aprotinin in Neonates Undergoing Cardiopulmonary Bypass: A Retrospective Chart Review
Brief Title: Aprotinin in Neonates Undergoing Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Angela Carrico, Mgr., Children's Healthcare of Atlanta Institutional Review Board
Other Study IDs: 07-020
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2010-05

CONDITIONS: Cardiopulmonary Bypass; Congenital Defects; Hemostasis
Keywords: Cardiology; Pediatrics; Cardiac Defects; Cardiopulmonary Bypass Surgery; Aprotinin; thrombosis; renal dysfunction
MeSH Terms: conditions — Congenital Abnormalities; Thrombosis; Renal Insufficiency

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective chart review study. The purpose of this study is to review our experience at Children's Healthcare of Atlanta in neonates receiving aprotinin. We will examine the specific outcomes of renal dysfunction, thrombosis and mortality.

DETAILED DESCRIPTION:
Aprotinin (Trasylol; Bayer Corporation, Pittsburgh, PA), a serine protease inhibitor isolated from bovine lung, is used intra-operatively during cardiac surgery to reduce bleeding. It is thought to work by inhibiting the contact activation phase of the coagulation cascade, reducing thrombin generation, preventing fibrinolysis and attenuating cardiopulmonary bypass (CPB)-induced platelet dysfunction.Though the efficacy of aprotinin in reducing blood loss in adults undergoing CPB is well established, its safety profile, specifically its association with renal dysfunction, thrombosis and long-term mortality, has been questioned. Although the homeostatic derangements of CPB are more significant in pediatric patients, its efficacy and safety profiles in this patient population are actually less clear. In children undergoing re-operative cardiac surgical procedures, aprotinin has been shown to be effective in attenuating post-bypass coagulopathies and decreasing blood product exposure (4). However, little information is available for neonates undergoing CPB who receive intra-operative aprotinin especially in terms of renal dysfunction and thrombosis.

All neonates who underwent Cardiopulmonary Bypass surgery (CPB) at Children's Healthcare of Atlanta between March 1, 2004 and March 1, 2007 will be candidates for this retrospective chart review. Notations will be made regarding those who received aprotinin and those who did not. Primary end points will include post-operative renal dysfunction, need for temporary dialysis, thrombosis and in-hospital mortality. Post -operative renal dysfunction will be defined as a doubling of the pre-operative creatinine level within the first 72 hours after surgery. Thrombosis found during the initial hospitalization will be considered significant. Chart review will gather demographic data (age, weight and type of surgery) as well as other data including CPB time, aortic cross clamp time, presence of regional perfusion, lowest temperature on CPB, time to chest closure, hours with a NIRS value below 40 in the first 24 hours post-op, highest recorded lactate value, blood products administered in the first 24 hours post-op, chest tube drainage in the first 24 hours post-op, first post-op weight, time to extubation and time to ICU discharge.

ELIGIBILITY:
Inclusion Criteria:

* Neonates who underwent Cardiopulmonary Bypass (CPB) at Children's Healthcare of Atlanta between March 2004 and March 2007.

Exclusion Criteria:

* All candidates who do not meet inclusion criteria.

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: neonates who underwent Cardiopulmonary Bypass (CPB) at Chldren's Healthcare of Atlanta between March 2004 and March 2007.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2007-04; Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Guzzetta, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Background] Dietrich W, Spath P, Zuhlsdorf M, Dalichau H, Kirchhoff PG, Kuppe H, Preiss DU, Mayer G. Anaphylactic reactions to aprotinin reexposure in cardiac surgery: relation to antiaprotinin immunoglobulin G and E antibodies. Anesthesiology. 2001 Jul;95(1):64-71; discussion 5A-6A. doi: 10.1097/00000542-200107000-00015. PMID 11465586
- [Background] Arnold DM, Fergusson DA, Chan AK, Cook RJ, Fraser GA, Lim W, Blajchman MA, Cook DJ. Avoiding transfusions in children undergoing cardiac surgery: a meta-analysis of randomized trials of aprotinin. Anesth Analg. 2006 Mar;102(3):731-7. doi: 10.1213/01.ane.0000194954.64293.61. PMID 16492820
- [Background] Mangano DT, Miao Y, Vuylsteke A, Tudor IC, Juneja R, Filipescu D, Hoeft A, Fontes ML, Hillel Z, Ott E, Titov T, Dietzel C, Levin J; Investigators of The Multicenter Study of Perioperative Ischemia Research Group; Ischemia Research and Education Foundation. Mortality associated with aprotinin during 5 years following coronary artery bypass graft surgery. JAMA. 2007 Feb 7;297(5):471-9. doi: 10.1001/jama.297.5.471. PMID 17284697
- [Background] Miller BE, Tosone SR, Tam VK, Kanter KR, Guzzetta NA, Bailey JM, Levy JH. Hematologic and economic impact of aprotinin in reoperative pediatric cardiac operations. Ann Thorac Surg. 1998 Aug;66(2):535-40; discussion 541. doi: 10.1016/s0003-4975(98)00469-x. PMID 9725399